CLINICAL TRIAL: NCT04868695
Title: Subjective and Objective Outcom Eof Endoscopic Sinus Surgery in Patients With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Subjective and Objective Outcome of ESS in CRSwNP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 2020-00322
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: CRS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bilateral Spheno-Ethmoidectomy: (Experimental)
  Interventions: Procedure: 1) Fronto-Sphenoethmoidektomie 2) Draf 2b 3) Draf 3
- Bilateral Fronto-Spheno-Ethmoidectomy + Draf 2b (Experimental)
  Interventions: Procedure: 1) Fronto-Sphenoethmoidektomie 2) Draf 2b 3) Draf 3
- Draf Typ 3 (Experimental)
  Interventions: Procedure: 1) Fronto-Sphenoethmoidektomie 2) Draf 2b 3) Draf 3

INTERVENTIONS:
Procedure: 1) Fronto-Sphenoethmoidektomie 2) Draf 2b 3) Draf 3 — 1) Fronto-Sphenoethmoidektomie 2) Draf 2b 3) Draf 3

SUMMARY:
(A): Beidseitige Fronto-Spheno-Ethmoidektomie mit Erweiterung des natürlichen Zuganges zur Stirnhöhle (Draf Typ II): Unter einem Draf Typ II Zugang versteht man die Erweiterung des natürlichen Zuganges zur Stirnhöhle mit Entfernung des Bodens der Stirnhöhle zwischen der Lamina papyracea zur Augenhöhle und der mittleren Nasenmuschel.

(B): Beidseitige Fronto-Spheno-Ethmoidektomie mit maximaler Erweiterung des Zuganges zur Stirnhöhle (Draf Typ III): Unter einem Draf Typ III verste. (C) Beidseitige Spheno-Ethmoidektomie: Abtragung des Processus uncinatus, die Eröffnung der Kieferhöhle, die Eröffnung des vorderen und hinteren Siebbeinsystems und die Eröffnung der Keilbeinhöhle.

DETAILED DESCRIPTION:
(A): Beidseitige Fronto-Spheno-Ethmoidektomie mit Erweiterung des natürlichen Zuganges zur Stirnhöhle (Draf Typ II): Unter einem Draf Typ II Zugang versteht man die Erweiterung des natürlichen Zuganges zur Stirnhöhle mit Entfernung des Bodens der Stirnhöhle zwischen der Lamina papyracea zur Augenhöhle und der mittleren Nasenmuschel.

(B): Beidseitige Fronto-Spheno-Ethmoidektomie mit maximaler Erweiterung des Zuganges zur Stirnhöhle (Draf Typ III): Unter einem Draf Typ III verste. (C) Beidseitige Spheno-Ethmoidektomie: Abtragung des Processus uncinatus, die Eröffnung der Kieferhöhle, die Eröffnung des vorderen und hinteren Siebbeinsystems und die Eröffnung der Keilbeinhöhle.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic CRSwNP patients without improvement after conservative treatment for at least 6 months Extent of disease at least Davos Polyp Score ≥ 4 points Age 18-65 years Signed consent

Exclusion Criteria:

* Previous sinunasal surgery High resolution paranasal sinus CT shows other pathology (e.g. mucocele) Incapable of judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyp Score | 12 months
  Nasal Polyps

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided